CLINICAL TRIAL: NCT03811522
Title: Comparison Air Versus Carbon Dioxide Insufflation in Single Balloon Anterograde Enteroscopy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: North Eastern Ohio Gastroenterology and Endoscopy center (Other)
Collaborators: Mercy Health Ohio (Other)
Responsible Party: Sponsor
Other Study IDs: NEOGastro
Record Dates: First submitted 2019-01-11; First posted 2019-01-22 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Carbon Dioxide Insufflation; Anterograde Single Balloon Enteroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Carbon Dioxide Insufflation: Received CO2 insufflation during procedure
  Interventions: Other: carbon dioxide insufflation
- Air Sufflation: Received ambient insufflation during procedure
  Interventions: Other: Air insufflation

INTERVENTIONS:
Other: carbon dioxide insufflation — Receives CO2 insufflation
  Groups: Carbon Dioxide Insufflation
Other: Air insufflation — Receives air insufflation
  Groups: Air Sufflation

SUMMARY:
Observation study comparing patient symptoms of bloating, pain, and nausea between CO2 insufflation vs. O2 insufflation in anterograde balloon enteroscopy.

DETAILED DESCRIPTION:
Study Subjects:

Patients >18 years of age who presented to North Eastern Ohio Gastroenterology and Associates and meet the indications for anterograde or retrograde balloon endoscopy. Indications include small intestinal bleeding, evaluation of small bowel mass, or evaluation and treatment of small bowel strictures. Patients excluded from the study are those who wish not to participate, pregnant patients, mentally disabled individuals, prisoners, patients who have long-term analgesic use (greater than 3 months) in the past 6 months from procedure date, or those patients deemed too high risk to undergo balloon endoscopy. High risk patients will be defined as have 3 or more of the following risk factors: chronic obstructive pulmonary disease, renal failure, morbid obesity (BMI > 40), immunosuppression, acquired/concurrent infection, diabetes, and chronic steroid use. Pre-operative risk will also be assessed by Dr. Dodig and GI fellow. ASA classifications will be evaluated on every patient by St. Joseph's staff anesthesiologist. Given that the patient is receiving general anesthesia, it is hospital policy that they are evaluated at the hospital by anesthesia team prior to the procedure for assessment of risk. Should a patient elect not to participate in the study they will receive the standard of care.

Subject Recruitment/Screening/Consent:

Patients will be recruited/consented/randomized by the GI fellow and advanced anterograde balloon endoscopist during the patient's routine office visit to discuss their pending procedure. This will take place in a private consultation room to ensure privacy and should take approximately 10-15 minutes. In order to minimize coercion, it will be made very clear to patients that their participation is voluntary and that participation will in no way affect their future care. Randomization will be performed using a sealed envelope system. All patients are to receive a copy of the informed consent.

Study Procedures:

The single balloon enteroscopy is performed with Olympus (SIF-Q180) and operated by a single experienced endoscopist, Dr. Milan Dodig, with over 1,000 single balloon endoscopies have been performed. Additional assistance provided via 3 gastroenterology fellows (Ryan Carbaugh D.O., Thomas Geisler D.O., and Justin Cochran D.O.). All anterograde enteroscopy procedures are to be performed in the surgical suite with general anesthesia. Patient CO2 levels will be non-invasively monitored by anesthesia with End-Tidal Carbon Dioxide (ETCO2). Anesthesia will be administered at the discretion of the consulting anesthesiologist via fentanyl, versed, and propofol. Insufflation utilized during procedure determined via randomization to air or carbon dioxide prior to procedure. The rate of air or carbon dioxide (level) is left to discretion of acting endoscopists for proper insufflation of bowel to achieve adequate luminal views. CO2 insufflator to be used is a Stratus CO2 insufflator made by Medivators.

After completion of procedure determination of patient pain level will be assessed at 15 minutes, 30 minutes, and 1-hour and 24-hour intervals using a patient survey. Pain is assessed based on the horizontal assessment scale (HAS). This scale based on a horizontal line measuring 100mm in length. Patient will be asked at the afore mentioned time intervals to mark with pen their level of pain on the HAS. The mark will then be measured in millimeters to determine score of pain. Score will be in a range from 0 to 100mm. Zero being no pain at all and 100mm the maximum pain level. The HAS is then documented with type of insufflation utilized and time interval. Patient will also be asked about nausea, abdominal fullness, and bloating after procedure to be ranked on a 0 to 10 scale, with zero being nothing to 10 as severe. This will also be ascertained at 15 minutes, 30 minutes, 1 hours and 24 hours. The 24 hours assessment for pain as well as dyspepsia symptoms is achieved through patients receiving HAS scale along with a questionnaire asking to rank dyspeptic symptoms. The HAS scale and dyspeptic questionnaire will be marked with patient identification number. A self-address envelope with postage will be given to patient with instruction return once completed within 24 hours of original procedure. Instruction sheets along with how to take dyspeptic survey will also be given.

Statistical Methods:

Data will be entered into Microsoft Excel 2017 and SPSS version 22 statistical programs. Analysis will include descriptive statistics, t-test, standard error, Pearson and fisher exact test. Statistical significance will be established with an alpha of 0.05 for all comparisons.

Adverse Events:

Risks consist of those entailed with general anesthesia and single balloon endoscopy.

The risk of CO2 insufflation consists of respiratory depression and CO2 embolism.16

Recording of Adverse Events:

At each contact with the subject, the investigator will seek information on adverse events by specific questioning and, as appropriate, by examination. Information on all adverse events will be recorded immediately (e.g., signs, symptoms, abnormal diagnostic procedures). The clinical course of each event will be followed until resolution, stabilization, or until it has been determined that the study treatment or participation is not the cause.

Reporting of Serious Adverse Events Reports of all serious adverse events (including follow-up information) will be submitted to the St. Elizabeth's Mercy Health IRB within five business days.

Data Management and Confidentiality Patient data will be entered into electronic spreadsheets. The spreadsheet will be stored as separate file, protected by unique passwords. Only the investigators will have access to the files and their passwords. Paper records will be stored in hard copy in a locked filing cabinet in the investigator's office or at the hospital's endoscopy suit. Should any new significant findings be made during the study, the patient will be made privy to these findings in a timely manner.

Provisions to Protect the Privacy Interests of Subjects Patient consent and all other research related activities will take place in a private exam room. Patient will also be receiving a copy of their informed consent.

Funding Source:

No funding is being sought for this study or being received.

ELIGIBILITY:
Inclusion Criteria:

* All patients who presented to North Eastern Ohio Gastroenterology and Associates and meet the indications for anterograde single balloon endoscopy. Indications include small intestinal bleeding, evaluation of small bowel mass, or evaluation and treatment of small bowel strictures.

Exclusion Criteria:

* Those who wish not to participate, pregnant patients, mentally disabled individuals, prisoners, patients who have long-term analgesic use (greater than 3 months) in the past 6 months from procedure date, or those patients deemed too high risk to undergo balloon endoscopy. High risk, defined as have 3 or more of the following risk factors: chronic obstructive pulmonary disease, renal failure, morbid obesity (BMI > 40), immuno-suppression, acquired/concurrent infection, diabetes, and chronic steroid use.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients >18 years of age who presented to North Eastern Ohio Gastroenterology and Associates and meet the indications for anterograde or retrograde balloon endoscopy. Indications include small intestinal bleeding, evaluation of small bowel mass, or evaluation and treatment of small bowel strictures. Patients excluded from the study are those who wish not to participate, pregnant patients, mentally disabled individuals, prisoners, patients who have long-term analgesic use (greater than 3 months) in the past 6 months from procedure date, or those patients deemed too high risk to undergo balloon endoscopy.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
The reduction of post operational pain | the survey will be asked at 15minutes, 30minutes, 1hour, and 24hours post op.
  Assessment of post operational pain will be made by the the horizontal assessment scale (HAS) for post operative pain. The survey will include the following questions.
  1. Mark your level of pain by drawing a horizontal line on the scale below.
  2. Rate the severity of your nausea by circling a number on the scale.
  3. Rate the severity of your bloating by circling a number on the scale.
  4. Rate the severity of your abdominal fullness by circling a number on the scale.
     * Note the scale was not provided given the limitation of characters.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Geisler, D.O., Principal Investigator — North Eastern Ohio Gastroenterology and Endoscopy center
Locations (1):
- St. Joesph Health Center, Warren, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sajid MS, Caswell J, Bhatti MI, Sains P, Baig MK, Miles WF. Carbon dioxide insufflation vs conventional air insufflation for colonoscopy: a systematic review and meta-analysis of published randomized controlled trials. Colorectal Dis. 2015 Feb;17(2):111-23. doi: 10.1111/codi.12837. PMID 25393051
- [Background] Fernandez-Calderon M, Munoz-Navas MA, Carrascosa-Gil J, Betes-Ibanez MT, de-la-Riva S, Prieto-de-Frias C, Herraiz-Bayod MT, Carretero-Ribon C. Carbon dioxide vs. air insufflation in ileo-colonoscopy and in gastroscopy plus ileo-colonoscopy: a comparative study. Rev Esp Enferm Dig. 2012 May;104(5):237-41. doi: 10.4321/s1130-01082012000500003. PMID 22662775
- [Background] ASGE Technology Committee; Lo SK, Fujii-Lau LL, Enestvedt BK, Hwang JH, Konda V, Manfredi MA, Maple JT, Murad FM, Pannala R, Woods KL, Banerjee S. The use of carbon dioxide in gastrointestinal endoscopy. Gastrointest Endosc. 2016 May;83(5):857-65. doi: 10.1016/j.gie.2016.01.046. Epub 2016 Mar 3. No abstract available. PMID 26946413
- [Background] Riverso M, Perbtani YB, Shuster JJD, Chakraborty J, Brar TS, Agarwal M, Zhang H, Gupte A, Chauhan SS, Forsmark CE, Draganov PV, Yang D. Carbon dioxide insufflation is associated with increased serrated polyp detection rate when compared to room air insufflation during screening colonoscopy. Endosc Int Open. 2017 Sep;5(9):E905-E912. doi: 10.1055/s-0043-116382. Epub 2017 Sep 13. PMID 28924598
- [Background] Yasumasa K, Nakajima K, Endo S, Ito T, Matsuda H, Nishida T. Carbon dioxide insufflation attenuates parietal blood flow obstruction in distended colon: potential advantages of carbon dioxide insufflated colonoscopy. Surg Endosc. 2006 Apr;20(4):587-94. doi: 10.1007/s00464-005-0252-0. Epub 2006 Jan 25. PMID 16437273
- [Background] Stavropoulos SN, Desilets DJ, Fuchs KH, Gostout CJ, Haber G, Inoue H, Kochman ML, Modayil R, Savides T, Scott DJ, Swanstrom LL, Vassiliou MC. Per-oral endoscopic myotomy white paper summary. Surg Endosc. 2014 Jul;28(7):2005-19. doi: 10.1007/s00464-014-3630-7. Epub 2014 Jun 17. No abstract available. PMID 24935204
- [Background] Navarro-Ripoll R, Martinez-Palli G, Guarner-Argente C, Cordova H, Martinez-Zamora MA, Comas J, Rodriguez de Miguel C, Beltran M, Rodriguez-D'Jesus A, Hernandez-Cera C, Llach J, Balust J, Fernandez-Esparrach G. On-demand endoscopic CO2 insufflation with feedback pressure regulation during natural orifice transluminal endoscopic surgery (NOTES) peritoneoscopy induces minimal hemodynamic and respiratory changes. Gastrointest Endosc. 2012 Aug;76(2):388-95. doi: 10.1016/j.gie.2011.10.015. PMID 22817790
- [Background] Li X, Zhao YJ, Dai J, Li XB, Xue HB, Zhang Y, Xiong GS, Ohtsuka K, Gao YJ, Liu Q, Song Y, Fang JY, Ge ZZ. Carbon dioxide insufflation improves the intubation depth and total enteroscopy rate in single-balloon enteroscopy: a randomised, controlled, double-blind trial. Gut. 2014 Oct;63(10):1560-5. doi: 10.1136/gutjnl-2013-306069. Epub 2014 Mar 13. PMID 24626435
- [Background] Lenz P, Meister T, Manno M, Pennazio M, Conigliaro R, Lebkucher S, Ullerich H, Schmedt A, Floer M, Beyna T, Lenze F, Domagk D. CO2 insufflation during single-balloon enteroscopy: a multicenter randomized controlled trial. Endoscopy. 2014 Jan;46(1):53-8. doi: 10.1055/s-0033-1359041. Epub 2013 Dec 18. PMID 24353124

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT03811522/Prot_SAP_003.pdf
  • Informed Consent Form (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT03811522/ICF_004.pdf